CLINICAL TRIAL: NCT01849380
Title: Neoadjuvant Epirubicin-cyclophosphamide-S-1 (ECS) Versus Epirubicin-cyclophosphamide-5-FU (ECF) in Local Advanced Breast Cancer
Brief Title: Neoadjuvant ECS Versus ECF in Local Advanced Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yu-Zhi Gang, Director of Department of Breast Disease, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEST T-01
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Breast Neoplasms; Neoadjuvant Therapy
Keywords: Local Advanced Breast Neoplasms; Neoadjuvant Chemotherapy; S-1
MeSH Terms: conditions — Breast Neoplasms | interventions — S 1 (combination); Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epirubicin-cyclophosphamide-S-1( ECS) (Experimental): S-1(SuLi,QILU Pharmaceutical co.ltd ) was given at a standard dose of 40 mg/m2 twice daily in cycles of 14-day consecutive administration followed by a 14-day rest, combined with by epirubicin(80mg/m2, d1 and d8 respectively) and cyclophosphamide(500mg/m2, d1, infusion). The chemotherapy was applicated 4 cycles 4-weekly.
  Interventions: Drug: S-1
- Epirubicin-cyclophosphamide-5-FU (ECF) (Active Comparator): 5-FU was given at a standard dose of 500mg/m2 (infusion, d1, d8 respectively), combined with by epirubicin(80mg/m2, d1 and d8 respectively) and cyclophosphamide(500mg/m2, d1, infusion). The chemotherapy was applicated 4 cycles 4-weekly.
  Interventions: Drug: 5-FU

INTERVENTIONS:
Drug: S-1 — S-1(SuLi, QILU Pharmaceutical co.ltd ) was given at a standard dose of 40 mg/m2 twice daily in cycles of 14-day consecutive administration
  Other Names: SuLi, QILU Pharmaceutical co.ltd
  Arms: Epirubicin-cyclophosphamide-S-1( ECS)
Drug: 5-FU — 5-FU was given at a standard dose of 500mg/m2 (infusion, d1, d8 respectively),
  Arms: Epirubicin-cyclophosphamide-5-FU (ECF)

SUMMARY:
S-1 is a newly developed novel oral dihydrouracil dehydrogenase inhibiting fluoro-pyrimidine drug consisting of i M tegafur (FT), 0.4 M 5-chloro-2, 4-dihydroxypyrimidine (gimeracil), and 1 M potassium oxonate (oteracil), with efficient antitumor activity and low gastrointestinal toxicity. Several studies have proved the safety and efficacy of single agent S-1 in metastatic breast cancer. This study is designed to further investigate and compare the efficacy and safety of Epirubicin-cyclophosphamide-S-1(ECS) vs. Epirubicin-cyclophosphamide-5-fluorouracil (ECF) as neoadjuvant chemotherapy in patients with local advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Disease characteristic:

  * Histologically confirmed primary breast cancer by core biopsy (Mammotome or bard needle)
  * Disease stage appropriate for neoadjuvant chemotherapy (T≥3cm, N0 or T（2-3cm）N1 or any T, N2)
  * Her-2(-); Ki67≥14%
  * No previous treatment for breast cancer (chemotherapy, endocrinotherapy, radiotherapy)
* Patients characteristic:

  * Female patients, age 18 to 70 years old
  * Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-2
  * Life expectancy of at least 12 weeks
  * Willing to be kept follow-up
  * Functions below are maintained in major organs:
  * Cardiac status:

LVEF: 50% 45% • Haematopoietic status: Leukocyte count: ≥4.0×109/L Neutrophil count: ≥2.0×109/L Platelet count: ≥100×109/L Hemoglobin: ≥80g/L

• Hepatic status: Total Bilirubin ≤ 1.5 x upper limit of normal (ULN), AST and ALT ≤ 2.5 times ULN(no liver metastasis) bilirubin:

• Renal status: BUN ≤ 1.5 x times ULN Creatinine ≤1.5 times ULN or calculated creatinine clearance, using the Cockcroft-Gault formula, ≥50 mL/min; Women's Ccr = Body weight x (140-Age)/(72 x Serum creatinine) x 0.85

• Written informed consent (both biopsy and neoadjuvant chemotherapy) will be obtained for patients for entering this study

Exclusion Criteria:

* Previous treatment for breast cancer (neither local nor systemic therapy)
* Known or suspected distant metastasis
* Potentially pregnant, pregnant, or breast-feeding
* Drug allergy
* Concurrent malignancy or history of other malignancy (except Hodgkin lymphoma)
* Currently active severe infection (Hepatitis included)
* History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures
* Known history of uncontrolled severe heart disease, myocardial infarction within 6 months, congestive heart failure, unstable angina pectoris, clinically significant hydropericardium or unstable arrhythmias

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-10 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 12 weeks
  Pathological complete response (pCR=ypT0 ypN0) rates of neoadjuvant treatment No microscopic evidence of residual invasive or non-invasive viable tumor cells in all resected specimens of the breast and axilla.
  Pathological response will be assessed considering all removed breast and lymphatic tissues from all surgeries.
  The primary endpoint will be summarized as pathological complete remission rate for each treatment group.
  Ultrasonic examination will be performed every 2 cycles of treatment for efficacy evaluation.

SECONDARY OUTCOMES:
Disease-free Survival | 5 years
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.
  Evaluation will be performed every 2 cycles of treatment during therapy, and follow-up will be performed every 3 months after therapy
Tolerability and safety | 12 weeks
  Reference to NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v 3.0. The endpoint will be summarized as events rate (%) for each treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Gang Z Yu, Dr; PhD, Principal Investigator — The Second Hospital of Shandong University
Locations (1):
- the Second Hospital of Shandong Universtity, Jinan, Shandong, China